CLINICAL TRIAL: NCT01891695
Title: A Pilot Single Arm Study of Intensity Modulated Radiation Therapy Elective Nodal Dose De-Escalation for HPV-Associated Squamous Cell Carcinoma of the Oropharynx
Brief Title: OPSCC N0 Nodal Control With Reduced IMRT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study had very specific inclusion/exclusion criteria and difficult to recruit
Sponsor: Paul W. Read, MD (Other)
Responsible Party: Sponsor-Investigator, Paul W. Read, MD, Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16766
Record Dates: First submitted 2013-06-24; First posted 2013-07-03 (Estimated); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma (OPSCCA); HPV (Human Papillomavirus)-Associated
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reduced Intensity Radiation (Experimental): 39.6 Gy radiation to clinically uninvolved cervical lymphatics
  Interventions: Radiation: 39.6 Gy radiation

INTERVENTIONS:
Radiation: 39.6 Gy radiation

SUMMARY:
The dose of radiation most commonly used to treat oropharyngeal cancer results in side effects including sores in the mouth and throat, dry mouth and thick saliva, loss or altered taste, swallowing problems including pain or inability to swallow requiring feeding tubes to be placed in the stomach, hoarseness or breathing problems from swelling requiring tracheostomy or a hole surgically placed in the windpipe to allow the patient to breathe, nausea and vomiting, fatigue and loss of energy, decreased hearing from fluid behind the ear drums in the middle ear, skin redness tenderness and blistering.

The purpose of this study is to determine if the investigators can reduce the dose of radiation to the lymph nodes in the neck that may contain cancer cells that are not detected by physical examinations or radiologic studies (CT scans, PET CT scans, or MRI scans) in order to reduce the side effects from treatment and still adequately kill any cancer cells that may be contained in those lymph nodes.

DETAILED DESCRIPTION:
A Pilot Single Arm Study of Intensity Modulated Radiation Therapy Elective Nodal Dose De-Escalation for HPV-Associated Squamous Cell Carcinoma of the Oropharynx.

ELIGIBILITY:
Inclusion Criteria:

* patient must be clinically referred for radiation for stage I-IVb OPSCCA
* tumor must be HPV-associated p16+
* patient must be able to lie flat and tolerate immobilization systems

Exclusion Criteria:

* patients may not be receiving any investigational agents
* prior radiation to head and neck
* any other malignancy except non-melanomatous skin cancer or a carcinoma not of head and neck origin with patient being disease free for at least 5 years
* any major medical, psychiatric, or neurologic illness
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Read, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced Intensity Radiation: 39.6 Gy radiation to clinically uninvolved cervical lymphatics
  39.6 Gy radiation
Period: Overall Study
Arm/Group | Reduced Intensity Radiation
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reduced Intensity Radiation
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 59 [59 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: N0 Nodal Control Rate
Description: Effectiveness of 39.6 Gy (Gray) radiation on tumor control in the clinically uninvolved (N0) cervical lymphatics of patients with p16+ oropharyngeal squamous cell carcinoma (OPSCCA)
Time Frame: Up to 3 years post treatment
Population: Study was stopped prematurely after 1 subject was enrolled. No analysis was performed.
Arm/Group | Reduced Intensity Radiation
Number analyzed (Participants) | 0

2. Secondary Outcome: Adverse Events of Participants Treated With 39.6 Gy Radiation to the Clinically Uninvolved Neck
Description: Evaluated safety and tolerability of treatment of p16+ OPSCCA by overall incidence of adverse events, incidence of acute and late toxicities and subject-rated quality of life assessments.
Time Frame: Up to 3 years post treatment
Population: Study was terminated after one subject enrolled. No analysis performed.
Arm/Group | Reduced Intensity Radiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival Following 39.6 Gy Radiation to the Clinically Uninvolved Neck
Description: Patient status reviewed and confirmed through Neck CT and PET scans at follow up time points throughout trial
Time Frame: Up to 3 years post treatment
Population: No analysis performed. Study was terminated after one subject was enrolled.
Arm/Group | Reduced Intensity Radiation
Number analyzed (Participants) | 0

4. Secondary Outcome: Dose Volume Histograms (DVH)
Description: Comparison of DVH of treatment plans between patients receiving 39.6 Gy versus the standard dose of 50 Gy to the clinically uninvolved neck
Time Frame: Up to 3 years post treatment
Population: Study was halted early. Only one subject was enrolled. No analysis performed.
Arm/Group | Reduced Intensity Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Reduced Intensity Radiation
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Intensity Radiation (N=1)
depression (Psychiatric disorders) | 1 (1)
Myelitis (Infections and infestations) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspahgiz (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
WBC decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Small intestine obstruction (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-04-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT01891695/Prot_SAP_000.pdf
  • Informed Consent Form (2013-06-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT01891695/ICF_001.pdf